CLINICAL TRIAL: NCT02570152
Title: A Cohort Study to Determine the Incidence of Dengue Fever and to Build Capacity for Dengue Vaccine Trials in Dengue-endemic Regions of South Asia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Ministry of Health, Sri Lanka (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200274
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Dengue
Keywords: Dengue; Non-laboratory confirmed dengue (non-LCD); Acute febrile illness (AFI); Laboratory confirmed dengue (LCD)
MeSH Terms: conditions — Dengue

ARMS (1):
- AFI Group (Experimental): Population living in randomly selected households in geographically-defined communities. Households including at least one member aged less than 18 years will be considered eligible if at least one adult (aged no more than 50 years) and one child (aged less than 18 years) consent (and assent if applicable) to participate in the study.
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — Blood samples will be collected during the Suspected Dengue First Visit. All study subjects with AFI (fever [body temperature ≥ 38°C/≥ 100.4°F] on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart) should be seen at a designated study hospital/clinic by the study physician. The Suspected Dengue First Visit should be scheduled within 7 days from the onset of fever (Days 2-7) and should ideally take place on the second day of fever (Day 2).

SUMMARY:
The purpose of this study is to determine the incidence of dengue fever and to build capacity for dengue vaccine trials in dengue-endemic regions of South Asia.

DETAILED DESCRIPTION:
This study aims to estimate the burden of dengue illness in selected sites South Asia and to prepare sites for the conduct of future vaccine efficacy trials.

Operational goals include:

* Build long-term collaboration with sites in dengue-endemic regions of South Asia where the incidence of clinical dengue illness can be studied.
* Establish dengue surveillance cohorts that can be followed long-term.
* Establish operational feasibility of future Phase III studies with regard to recruitment, case capture and sampling procedures.
* Prepare sites for participation in Phase III clinical endpoint studies.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's parent(s)/legally acceptable representative(s) (LAR[s]) who, in the opinion of the investigator, can and will comply with the requirements of the protocol. (e.g., willingness to go to the hospital/clinic for visit[s] in case of AFI, able to observe the signs of dengue and to understand how to take and report body temperature, etc.).
* Signed/thumb-printed (and video recorded if required by law) informed consent (and assent if applicable) must be obtained from the subject/subject's parent(s)/LAR(s) at the hospital/clinic or during a home visit. If the subject/subject's parent(s)/LAR(s) are illiterate, the informed consent form (ICF) (or informed assent form [IAF] when applicable) will be countersigned by an impartial witness.
* Subject is part of a household with at least one child (aged less than 18 years) and in which informed consent (and assent if applicable) to study participation was obtained from at least one adult and one child.
* Male or female aged between and including 6 months and 50 years at the time of enrolment.
* Subject who plans, at the time of enrolment, to remain at same residence/study area during the two-year study period.

Exclusion Criteria:

* Child in care.
* Participation (current or planned) in another epidemiological study or in a clinical trial that would conflict with the current study, based on investigator's judgement.
* Terminal illness based on investigator's judgement.
* Mental incapacity based on investigator's judgement.

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2004 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Colombo, Sri Lanka

REFERENCES:
- [Derived] Tissera H, Samaraweera P, de Boer M, Gandhi S, Malvaux L, Mehta S, Palihawadana P, Vantomme V, Paris R, Schmidt A. The Burden of Acute Febrile Illness Attributable to Dengue Virus Infection in Sri Lanka: A Single-Center 2-Year Prospective Cohort Study (2016-2019). Am J Trop Med Hyg. 2021 Nov 1;106(1):160-167. doi: 10.4269/ajtmh.21-0604. PMID 34724624

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Subjects aged between 6 months and 50 years at the time of enrollment, living in randomly selected households in geographically-defined communities. Households including at least one member aged less than 18 years were considered eligible if at least one adult (aged no more than 50 years) and one child (aged less than 18 years) consented (and assented if applicable) to participate in the study.
Period: Overall Study
Arm/Group | Study Group
Started (2004) | 2004
Completed (1989) | 1989
Not Completed | 15
Not completed — Protocol Violation | 2
Not completed — Migrated/moved from study area | 13

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1038
  Male | 966
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Laboratory Confirmed Dengue (LCD) Overall, and by Age Group
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to LCD) OR date of last contact OR date of death. An AFI due to LCD was confirmed if all of the following criteria were met: Fever (body temperature greater than or equal to (≥) 38°Celsius [C]/≥ 100.4°Farhenheit [F] on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart AND Laboratory confirmation of dengue through dengue Reverse Transcriptase quantitative Polymerase Chain Reaction (RT-qPCR) on acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F).
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Person-year rate ( Per 1000)
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Person-year rate ( Per 1000)
  <5 years: number analyzed (Participants) | 257
  <5 years | 21.25 [10.61 to 38.02]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 22.69 [13.66 to 35.44]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 12.76 [5.13 to 26.3]
  ≥ 18 years: number analyzed (Participants) | 1033
  ≥ 18 years | 9.16 [5.43 to 14.47]
  Overall | 14.21 [10.71 to 18.5]

2. Secondary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Non-Laboratory Confirmed Dengue (Non-LCD) Overall, and by Age Group
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to non-LCD) OR date of last contact OR date of death. An AFI due to non-LCD was confirmed if all of the following criteria were met: Fever (body temperature ≥ 38°C/≥ 100.4°F) on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart, AND Dengue RT-qPCR result on the acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F) was (valid but) negative for dengue.
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-year
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Events per 1000 person-year
  <5 years: number analyzed (Participants) | 257
  <5 years | 104.31 [78.36 to 136.11]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 84.8 [66.23 to 106.97]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 43.76 [28.04 to 65.11]
  ≥ 18 years: number analyzed (Participants) | 1033
  ≥ 18 years | 17.3 [11.98 to 24.17]
  Overall | 47.3 [40.69 to 54.67]

3. Secondary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Laboratory Confirmed Sero Type 1 Dengue Overall, and by Age Group.
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to LCD Sero Type 1) OR date of last contact OR date of death. An AFI due to LCD Sero Type 1 was confirmed if all of the following criteria were met: Fever (body temperature greater than or equal to (≥) 38°C/≥ 100.4°F on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart AND Laboratory confirmation of dengue Sero Type 1 through RT-qPCR on acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F).
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-year
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Events per 1000 person-year
  <5 years: number analyzed (Participants) | 257
  <5 years | 0 [0 to 7.13]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 3.59 [0.74 to 10.48]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 0 [0 to 6.73]
  ≥ 18: number analyzed (Participants) | 1033
  ≥ 18 | 1.53 [0.31 to 4.46]
  Overall | 1.55 [0.57 to 3.38]

4. Secondary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Laboratory Confirmed Sero Type 2 Dengue Overall, and by Age Group
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to LCD Sero Type 2) OR date of last contact OR date of death. An AFI due to LCD Sero Type 2 was confirmed if all of the following criteria were met: Fever (body temperature greater than or equal to (≥) 38°C/≥ 100.4°F on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart AND Laboratory confirmation of dengue Sero Type 2 through RT-qPCR on acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F).
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-year
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Events per 1000 person-year
  <5 years: number analyzed (Participants) | 257
  <5 years | 21.25 [10.61 to 38.02]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 17.94 [10.04 to 29.58]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 12.76 [5.13 to 26.3]
  ≥ 18 years: number analyzed (Participants) | 1033
  ≥ 18 years | 6.61 [3.52 to 11.31]
  Overall | 11.89 [8.71 to 15.86]

5. Secondary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Laboratory Confirmed Sero Type 3 Dengue Overall, and by Age Group
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to LCD Sero Type 3) OR date of last contact OR date of death. An AFI due to LCD Sero Type 3 was confirmed if all of the following criteria were met: Fever (body temperature greater than or equal to (≥) 38°C/≥ 100.4°F on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart AND Laboratory confirmation of dengue Sero Type 3 through RT-qPCR on acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F)
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-year
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Events per 1000 person-year
  <5 years: number analyzed (Participants) | 257
  <5 years | 0 [0 to 7.13]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 1.2 [0.03 to 6.66]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 0 [0 to 6.73]
  ≥ 18: number analyzed (Participants) | 1033
  ≥ 18 | 1.02 [0.12 to 3.68]
  Overall | 0.78 [0.16 to 2.27]

6. Secondary Outcome: Incidence Rate of Acute Febrile Illness (AFI) Due to Laboratory Confirmed Sero Type 4 Dengue Overall, and by Age Group
Description: The incidence rate of first event (IR per 1000 person-years) was calculated by dividing the number of subjects reporting at least one episode of event during the follow-up period by the total person-year at risk. The person-time at risk for an event of interest was calculated as the duration between the date of enrolment and the end of the at-risk period or the earliest of the following: onset date of event of interest (e.g. first episode of AFI due to LCD Sero Type 4) OR date of last contact OR date of death. An AFI due to LCD Sero Type 4 was confirmed if all of the following criteria were met: Fever (body temperature greater than or equal to (≥) 38°C/≥ 100.4°F on ≥ 2 consecutive calendar days, measured at least twice, at least 8 hours apart AND Laboratory confirmation of dengue Sero Type 4 through RT-qPCR on acute serum sample taken during the 7-day period (Days 2-7) from the onset of fever (body temperature ≥ 38°C/≥ 100.4°F)
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-year
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Events per 1000 person-year
  <5 years: number analyzed (Participants) | 257
  <5 years | 0 [0 to 7.13]
  5 to 11 years: number analyzed (Participants) | 433
  5 to 11 years | 0 [0 to 4.41]
  12 to 17 years: number analyzed (Participants) | 281
  12 to 17 years | 0 [0 to 6.73]
  ≥ 18: number analyzed (Participants) | 1033
  ≥ 18 | 0 [0 to 1.88]
  Overall | 0 [0 to 0.95]

7. Secondary Outcome: Number of Acute Febrile Illness Due to Laboratory Confirmed Dengue Presenting a Sign or a Symptom of Interest (Any Intensity) During the 7-day Period Following the Onset of Each Episode of AFI Due to LCD.
Description: Description of signs and symptoms of AFI due to LCD included the percentage of AFI presenting each sign or symptom (any intensity) during the 7-day period from the onset of fever (body temperature 38°C/100.4°F).
Time Frame: At each day during the 7-day period following the onset of each episode of AFI due to LCD
Population: Analysis was performed on all subjects enrolled in the study and with AFI due to LCD.
Measure: Count of Units; unit: AFI episodes
Units Other Than Participants: AFI episodes
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Number analyzed (AFI episodes) | 55
AFI episodes
  Headache / irritability at Day 1 | 51
  Headache / irritability at Day 2 | 51
  Headache / irritability at Day 3 | 51
  Headache / irritability at Day 4 | 51
  Headache / irritability at Day 5 | 51
  Headache / irritability at Day 6 | 50
  Headache / irritability at Day 7 | 50
  Eye pain at Day 1 | 34
  Eye pain at Day 2 | 34
  Eye pain at Day 3 | 34
  Eye pain at Day 4 | 34
  Eye pain at Day 5 | 34
  Eye pain at Day 6 | 34
  Eye pain at Day 7 | 34
  Myalgia (muscle pain) at Day 1 | 47
  Myalgia (muscle pain) at Day 2 | 47
  Myalgia (muscle pain) at Day 3 | 47
  Myalgia (muscle pain) at Day 4 | 47
  Myalgia (muscle pain) at Day 5 | 47
  Myalgia (muscle pain) at Day 6 | 47
  Myalgia (muscle pain) at Day 7 | 47
  Arthralgia (joint pain) at Day 1 | 42
  Arthralgia (joint pain) at Day 2 | 42
  Arthralgia (joint pain) at Day 3 | 42
  Arthralgia (joint pain) at Day 4 | 42
  Arthralgia (joint pain) at Day 5 | 42
  Arthralgia (joint pain) at Day 6 | 42
  Arthralgia (joint pain) at Day 7 | 42
  Abdominal pain at Day 1 | 31
  Abdominal pain at Day 2 | 31
  Abdominal pain at Day 3 | 31
  Abdominal pain at Day 4 | 31
  Abdominal pain at Day 5 | 31
  Abdominal pain at Day 6 | 31
  Abdominal pain at Day 7 | 31
  Nausea at Day 1 | 29
  Nausea at Day 2 | 29
  Nausea at Day 3 | 29
  Nausea at Day 4 | 29
  Nausea at Day 5 | 29
  Nausea at Day 6 | 29
  Nausea at Day 7 | 29
  Vomiting at Day 1 | 29
  Vomiting at Day 2 | 29
  Vomiting at Day 3 | 29
  Vomiting at Day 4 | 29
  Vomiting at Day 5 | 29
  Vomiting at Day 6 | 29
  Vomiting at Day 7 | 29
  Rash at Day 1 | 5
  Rash at Day 2 | 5
  Rash at Day 3 | 5
  Rash at Day 4 | 5
  Rash at Day 5 | 5
  Rash at Day 6 | 5
  Rash at Day 7 | 5
  Any bleeding (skin, mouth, anus) at Day 1 | 4
  Any bleeding (skin, mouth, anus) at Day 2 | 4
  Any bleeding (skin, mouth, anus) at Day 3 | 4
  Any bleeding (skin, mouth, anus) at Day 4 | 4
  Any bleeding (skin, mouth, anus) at Day 5 | 4
  Any bleeding (skin, mouth, anus) at Day 6 | 4
  Any bleeding (skin, mouth, anus) at Day 7 | 4
  Loss of appetite at Day 1 | 43
  Loss of appetite at Day 2 | 43
  Loss of appetite at Day 3 | 43
  Loss of appetite at Day 4 | 43
  Loss of appetite at Day 5 | 43
  Loss of appetite at Day 6 | 43
  Loss of appetite at Day 7 | 43
  Fatigue/decrease in normal activity at Day 1 | 48
  Fatigue/decrease in normal activity at Day 2 | 48
  Fatigue/decrease in normal activity at Day 3 | 48
  Fatigue/decrease in normal activity at Day 4 | 48
  Fatigue/decrease in normal activity at Day 5 | 48
  Fatigue/decrease in normal activity at Day 6 | 48
  Fatigue/decrease in normal activity at Day 7 | 48
  Reduced fluid intake at Day 1 | 33
  Reduced fluid intake at Day 2 | 33
  Reduced fluid intake at Day 3 | 33
  Reduced fluid intake at Day 4 | 33
  Reduced fluid intake at Day 5 | 33
  Reduced fluid intake at Day 6 | 33
  Reduced fluid intake at Day 7 | 33

8. Secondary Outcome: Number of Acute Febrile Illness Due to Laboratory Confirmed Dengue Presenting a Sign or a Symptom of Interest (Grade 3) During the 7-day Period Following the Onset of Each Episode of AFI Due to LCD
Description: Description of signs and symptoms of AFI due to LCD included the percentage of AFI presenting each sign or symptom (grade 3) during the 7-day period from the onset of fever (body temperature 38°C/100.4°F).
Time Frame: At each day during the 7-day period following the onset of each episode of AFI due to LCD
Population: Analysis was performed on all subjects enrolled in the study and with AFI due to LCD.
Measure: Count of Units; unit: AFI episodes
Units Other Than Participants: AFI episodes
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Number analyzed (AFI episodes) | 55
AFI episodes
  Headache / irritability at Day 1 | 11
  Headache / irritability at Day 2 | 11
  Headache / irritability at Day 3 | 11
  Headache / irritability at Day 4 | 11
  Headache / irritability at Day 5 | 11
  Headache / irritability at Day 6 | 11
  Headache / irritability at Day 7 | 11
  Eye pain at Day 1 | 2
  Eye pain at Day 2 | 2
  Eye pain at Day 3 | 2
  Eye pain at Day 4 | 2
  Eye pain at Day 5 | 2
  Eye pain at Day 6 | 2
  Eye pain at Day 7 | 2
  Myalgia (muscle pain) at Day 1 | 10
  Myalgia (muscle pain) at Day 2 | 10
  Myalgia (muscle pain) at Day 3 | 10
  Myalgia (muscle pain) at Day 4 | 10
  Myalgia (muscle pain) at Day 5 | 10
  Myalgia (muscle pain) at Day 6 | 10
  Myalgia (muscle pain) at Day 7 | 10
  Arthralgia (joint pain) at Day 1 | 8
  Arthralgia (joint pain) at Day 2 | 8
  Arthralgia (joint pain) at Day 3 | 8
  Arthralgia (joint pain) at Day 4 | 8
  Arthralgia (joint pain) at Day 5 | 8
  Arthralgia (joint pain) at Day 6 | 8
  Arthralgia (joint pain) at Day 7 | 8
  Abdominal pain at Day 1 | 2
  Abdominal pain at Day 2 | 2
  Abdominal pain at Day 3 | 2
  Abdominal pain at Day 4 | 2
  Abdominal pain at Day 5 | 2
  Abdominal pain at Day 6 | 2
  Abdominal pain at Day 7 | 2
  Vomiting at Day 1 | 1
  Vomiting at Day 2 | 1
  Vomiting at Day 3 | 1
  Vomiting at Day 4 | 1
  Vomiting at Day 5 | 1
  Vomiting at Day 6 | 1
  Vomiting at Day 7 | 1
  Rash at Day 1 | 1
  Rash at Day 2 | 1
  Rash at Day 3 | 1
  Rash at Day 4 | 1
  Rash at Day 5 | 1
  Rash at Day 6 | 1
  Rash at Day 7 | 1
  Loss of appetite at Day 1 | 8
  Loss of appetite at Day 2 | 8
  Loss of appetite at Day 3 | 8
  Loss of appetite at Day 4 | 8
  Loss of appetite at Day 5 | 8
  Loss of appetite at Day 6 | 8
  Loss of appetite at Day 7 | 8
  Fatigue/decrease in normal activity at Day 1 | 14
  Fatigue/decrease in normal activity at Day 2 | 14
  Fatigue/decrease in normal activity at Day 3 | 14
  Fatigue/decrease in normal activity at Day 4 | 14
  Fatigue/decrease in normal activity at Day 5 | 14
  Fatigue/decrease in normal activity at Day 6 | 14
  Fatigue/decrease in normal activity at Day 7 | 14
  Reduced fluid intake at Day 1 | 4
  Reduced fluid intake at Day 2 | 4
  Reduced fluid intake at Day 3 | 4
  Reduced fluid intake at Day 4 | 4
  Reduced fluid intake at Day 5 | 4
  Reduced fluid intake at Day 6 | 4
  Reduced fluid intake at Day 7 | 4

9. Secondary Outcome: Number of Acute Febrile Illness Due to Non-Laboratory Confirmed Dengue Presenting a Sign or a Symptom of Interest (Any Intensity) During the 7-day Period Following the Onset of Each Episode of AFI Due to Non-LCD
Description: Description of signs and symptoms of AFI due to non-LCD included the percentage of AFI presenting each sign or symptom (any intensity) during the 7-day period from the onset of fever (body temperature 38°C/100.4°F).
Time Frame: At each day during the 7-day period following the onset of each episode of AFI due to non-LCD
Population: Analysis was performed on all subjects enrolled in the study and with AFI due to non-LCD.
Measure: Count of Units; unit: AFI episodes
Units Other Than Participants: AFI episodes
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Number analyzed (AFI episodes) | 183
AFI episodes
  Headache / irritability at Day 1 | 159
  Headache / irritability at Day 2 | 159
  Headache / irritability at Day 3 | 159
  Headache / irritability at Day 4 | 157
  Headache / irritability at Day 5 | 158
  Headache / irritability at Day 6 | 158
  Headache / irritability at Day 7 | 158
  Eye pain at Day 1 | 80
  Eye pain at Day 2 | 80
  Eye pain at Day 3 | 80
  Eye pain at Day 4 | 78
  Eye pain at Day 5 | 79
  Eye pain at Day 6 | 79
  Eye pain at Day 7 | 78
  Myalgia (muscle pain) at Day 1 | 133
  Myalgia (muscle pain) at Day 2 | 133
  Myalgia (muscle pain) at Day 3 | 133
  Myalgia (muscle pain) at Day 4 | 131
  Myalgia (muscle pain) at Day 5 | 132
  Myalgia (muscle pain) at Day 6 | 132
  Myalgia (muscle pain) at Day 7 | 132
  Arthralgia (joint pain at Day 1 | 118
  Arthralgia (joint pain at Day 2 | 118
  Arthralgia (joint pain at Day 3 | 118
  Arthralgia (joint pain at Day 4 | 116
  Arthralgia (joint pain at Day 5 | 117
  Arthralgia (joint pain at Day 6 | 117
  Arthralgia (joint pain at Day 7 | 117
  Abdominal pain at Day 1 | 87
  Abdominal pain at Day 2 | 87
  Abdominal pain at Day 3 | 87
  Abdominal pain at Day 4 | 86
  Abdominal pain at Day 5 | 87
  Abdominal pain at Day 6 | 87
  Abdominal pain at Day 7 | 87
  Nausea at Day 1 | 92
  Nausea at Day 2 | 92
  Nausea at Day 3 | 92
  Nausea at Day 4 | 90
  Nausea at Day 5 | 91
  Nausea at Day 6 | 91
  Nausea at Day 7 | 91
  Vomiting at Day 1 | 71
  Vomiting at Day 2 | 71
  Vomiting at Day 3 | 71
  Vomiting at Day 4 | 70
  Vomiting at Day 5 | 71
  Vomiting at Day 6 | 71
  Vomiting at Day 7 | 71
  Rash at Day 1 | 7
  Rash at Day 2 | 7
  Rash at Day 3 | 7
  Rash at Day 4 | 7
  Rash at Day 5 | 7
  Rash at Day 6 | 7
  Rash at Day 7 | 7
  Any bleeding (skin, mouth, anus) at Day 1 | 6
  Any bleeding (skin, mouth, anus) at Day 2 | 6
  Any bleeding (skin, mouth, anus) at Day 3 | 6
  Any bleeding (skin, mouth, anus) at Day 4 | 6
  Any bleeding (skin, mouth, anus) at Day 5 | 6
  Any bleeding (skin, mouth, anus) at Day 6 | 6
  Any bleeding (skin, mouth, anus) at Day 7 | 6
  Loss of appetite at Day 1 | 140
  Loss of appetite at Day 2 | 140
  Loss of appetite at Day 3 | 140
  Loss of appetite at Day 4 | 138
  Loss of appetite at Day 5 | 139
  Loss of appetite at Day 6 | 139
  Loss of appetite at Day 7 | 137
  Fatigue/decrease in normal activity at Day 1 | 152
  Fatigue/decrease in normal activity at Day 2 | 152
  Fatigue/decrease in normal activity at Day 3 | 152
  Fatigue/decrease in normal activity at Day 4 | 150
  Fatigue/decrease in normal activity at Day 5 | 151
  Fatigue/decrease in normal activity at Day 6 | 151
  Fatigue/decrease in normal activity at Day 7 | 150
  Reduced fluid intake at Day 1 | 105
  Reduced fluid intake at Day 2 | 105
  Reduced fluid intake at Day 3 | 105
  Reduced fluid intake at Day 4 | 103
  Reduced fluid intake at Day 5 | 103
  Reduced fluid intake at Day 6 | 103
  Reduced fluid intake at Day 7 | 102

10. Secondary Outcome: Number of Acute Febrile Illness Due to Non-Laboratory Confirmed Dengue Presenting a Sign or a Symptom of Interest (Grade 3) During the 7-day Period Following the Onset of Each Episode of AFI Due to Non-LCD
Description: Description of signs and symptoms of AFI due to non-LCD included the percentage of AFI presenting each sign or symptom (grade 3) during the 7-day period from the onset of fever (body temperature 38°C/100.4°F).
Time Frame: At each day during the 7-day period following the onset of each episode of AFI due to non-LCD
Population: Analysis was performed on all subjects enrolled in the study and with AFI due to non-LCD.
Measure: Count of Units; unit: AFI episodes
Units Other Than Participants: AFI episodes
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Number analyzed (AFI episodes) | 183
AFI episodes
  Headache / irritability at Day 1 | 16
  Headache / irritability at Day 2 | 16
  Headache / irritability at Day 3 | 16
  Headache / irritability at Day 4 | 15
  Headache / irritability at Day 5 | 16
  Headache / irritability at Day 6 | 16
  Headache / irritability at Day 7 | 16
  Eye pain at Day 1 | 5
  Eye pain at Day 2 | 5
  Eye pain at Day 3 | 5
  Eye pain at Day 4 | 5
  Eye pain at Day 5 | 5
  Eye pain at Day 6 | 5
  Eye pain at Day 7 | 5
  Myalgia (muscle pain) at Day 1 | 14
  Myalgia (muscle pain) at Day 2 | 14
  Myalgia (muscle pain) at Day 3 | 14
  Myalgia (muscle pain) at Day 4 | 13
  Myalgia (muscle pain) at Day 5 | 14
  Myalgia (muscle pain) at Day 6 | 14
  Myalgia (muscle pain) at Day 7 | 14
  Arthralgia (joint pain) at Day 1 | 12
  Arthralgia (joint pain) at Day 2 | 12
  Arthralgia (joint pain) at Day 3 | 12
  Arthralgia (joint pain) at Day 4 | 11
  Arthralgia (joint pain) at Day 5 | 12
  Arthralgia (joint pain) at Day 6 | 12
  Arthralgia (joint pain) at Day 7 | 12
  Abdominal pain at Day 1 | 4
  Abdominal pain at Day 2 | 4
  Abdominal pain at Day 3 | 4
  Abdominal pain at Day 4 | 3
  Abdominal pain at Day 5 | 4
  Abdominal pain at Day 6 | 4
  Abdominal pain at Day 7 | 4
  Nausea at Day 1 | 4
  Nausea at Day 2 | 4
  Nausea at Day 3 | 4
  Nausea at Day 4 | 3
  Nausea at Day 5 | 4
  Nausea at Day 6 | 4
  Nausea at Day 7 | 4
  Vomiting at Day 1 | 4
  Vomiting at Day 2 | 4
  Vomiting at Day 3 | 4
  Vomiting at Day 4 | 3
  Vomiting at Day 5 | 4
  Vomiting at Day 6 | 4
  Vomiting at Day 7 | 4
  Rash at Day 1 | 1
  Rash at Day 2 | 1
  Rash at Day 3 | 1
  Rash at Day 4 | 1
  Rash at Day 5 | 1
  Rash at Day 6 | 1
  Rash at Day 7 | 1
  Loss of appetite at Day 1 | 11
  Loss of appetite at Day 2 | 11
  Loss of appetite at Day 3 | 11
  Loss of appetite at Day 4 | 11
  Loss of appetite at Day 5 | 11
  Loss of appetite at Day 6 | 11
  Loss of appetite at Day 7 | 11
  Fatigue/decrease in normal activity at Day 1 | 17
  Fatigue/decrease in normal activity at Day 2 | 17
  Fatigue/decrease in normal activity at Day 3 | 17
  Fatigue/decrease in normal activity at Day 4 | 16
  Fatigue/decrease in normal activity at Day 5 | 17
  Fatigue/decrease in normal activity at Day 6 | 17
  Fatigue/decrease in normal activity at Day 7 | 17
  Reduced fluid intake at Day 1 | 5
  Reduced fluid intake at Day 2 | 5
  Reduced fluid intake at Day 3 | 5
  Reduced fluid intake at Day 4 | 5
  Reduced fluid intake at Day 5 | 5
  Reduced fluid intake at Day 6 | 5
  Reduced fluid intake at Day 7 | 5

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to a Study Procedure
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first visit to last visit (approximatively 2 years per subject)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 2004
Participants | 0

ADVERSE EVENTS:
Time Frame: Any signs or symptoms were collected during the 7-day period following the onset of fever. Serious adverse events were collected from first visit to last visit (approximately 2 years per subject).
Description: The signs or symptoms collected were specified in the protocol and were not classified per MedDRA dictionary.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/2004
Serious Adverse Events (participants affected / at risk) | 0/2004
Other Adverse Events (participants affected / at risk) | 216/2004
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=2004)
Abdominal pain (General disorders) | 109 (109)
Arthralgia (General disorders) | 147 (147)
Bleeding (General disorders) | 10 (10)
Eye pain (General disorders) | 106 (106)
Fatigue (General disorders) | 186 (186)
Headache (General disorders) | 192 (192)
Loss of appetite (General disorders) | 170 (170)
Loss of appetite (General disorders) | 166 (166)
Nausea (General disorders) | 113 (113)
Rash (General disorders) | 11 (11)
Reduced fluid intake (General disorders) | 128 (128)
Vomiting (General disorders) | 99 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02570152/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT02570152/SAP_001.pdf